CLINICAL TRIAL: NCT04211350
Title: A Multi-center, Prospective, Randomized Crossover Study With the NightBalance SPT Compared to Positive Airway Pressure (PAP) for the Treatment of Positional Obstructive Sleep Apnea (POSA)
Brief Title: SLEEP ON Your SIDE (SOS) Study
Acronym: SOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Global recall of the comparator device
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EU-2018-001; 2018-A02141-54 (Other: CA ANSM (Agence nationale de sécurité du médicament et des produits de santé)); ISRCTN16170657 (Registry Identifier: ISRCTN registry)
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Positional Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NightBalance Sleep Position Therapy (Experimental): NightBalance Sleep Position Trainer (SPT) avoids POSA patients from sleeping on their back by delivering a vibrational stimulus, via a small device which is worn in a chest strap during sleep, each time the patient rolls to their back. This prompts the patient to roll over onto their side.
  Interventions: Device: NightBalance Sleep Position Trainer (SPT)
- Positive Airway Pressure (APAP) (Experimental): Automatic Positive Airway Pressure (APAP) is a pump that provides a positive flow of air to keep the airway open.
  Interventions: Device: Automatic Positive Airway Pressure (APAP)

INTERVENTIONS:
Device: NightBalance Sleep Position Trainer (SPT) — NightBalance Sleep Position Trainer (SPT) avoids POSA patients from sleeping on their back by delivering a vibrational stimulus, via a small device which is worn in a chest strap during sleep, each time the patient rolls to their back. This prompts the patient to roll over onto their side.
  Arms: NightBalance Sleep Position Therapy
Device: Automatic Positive Airway Pressure (APAP) — Automatic Positive Airway Pressure (APAP) is a pump that provides a positive flow of air to keep the airway open.
  Arms: Positive Airway Pressure (APAP)

SUMMARY:
Comparison of the NightBalance Sleep Position Trainer (SPT) to Positive Airway Pressure (PAP) for the Treatment of Positional Obstructive Sleep Apnea (POSA). Primary Objective: Efficacy and Adherence of the SPT over 3 months of use compared to PAP for the treatment of POSA. The study is run from centers in France, the UK and Germany.

DETAILED DESCRIPTION:
Participants are randomly allocated to receive one of two treatments, either Automatic Positive Airway Pressure (APAP) or NightBalance Sleep Position Therapy for a three month period. Participants are sent home with instructions to use that device nightly at home for three months. After three months of using the first device, they return to the doctor for assessment of the efficacy of the device using a sleep test and the compliance read from the device. Upon conclusion of the first three month treatment period, patients receive the alternative treatment for a further three months. At the end of the second three month period, participants return to their doctor again to assess the efficacy of the last device and read the compliance. Before any treatment and after each treatment, patients undergo a sleep test and complete some questionnaires. During each treatment period, patients complete a healthcare utilization diary and report any problems.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is adult
2. Either: Treatment naïve, or PAP non-complier (defined as current AAP user with <3 hours per night in the last 3 months per compliance download), and willing to use the APAP device per protocol
3. Diagnosis of POSA meeting all the following criteria per control PSG within 6 months of screening: AHI of >15 during PSG with symptoms of sleepiness per Investigator discretion, or AHI of >15 during respiratory polygraphy with comorbidities (e.g. atrial fibrillation, resistant hypertension, etc.)
4. Supine AHI at least twice the lateral AHI
5. Lateral AHI <10
6. Supine time >30% and <70%
7. Understands the study protocol and is willing and able to comply with study requirements and sign informed consent. APAP non-compliant subjects must be willing to use their APAP device per protocol.

Exclusion Criteria:

1. Prior or current therapy or treatment for OSA (for Treatment naïve group); Greater than an average of 3 hours per night of APAP use (in the APAP non-complier group)
2. A female of child-bearing potential that is pregnant or intends to become pregnant
3. Any unstable or severe medical condition of any organ system that at the discretion of the site Principal Investigator (PI) might affect the patient's participation in the study or generalization of treatment results
4. Taking medication that at the discretion of the site Principal Investigator (PI) might affect the patient's participation in the study or generalization of treatment results
5. Oxygen use
6. The presence of any other sleep disorder (central sleep apnea (CSA >5), periodic limb movement disorder (PLMAI >15), clinical diagnosis of insomnia or narcolepsy)
7. Excessive alcohol consumption (>21 drinks/week)
8. The use of any illegal drug(s), per subject report
9. Night or rotating shift work
10. Severe claustrophobia
11. Shoulder, neck, or back complaints that restrict sleeping position
12. Subject requires use of more than 2 pillows under the head while sleeping or sleeps in a bed/chair with raised upper body position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change of Apnea-Hypopnea Index (AHI) | Baseline,3 months and 6 months
  Efficacy will be measured as Change of Apnea-Hypopnea Index (AHI) from baseline to 3 months and from 3 months to 6 months (NightBalance SPT non-inferior to PAP)
Difference of the total hours medical device use between each treatment arm | 3 months and 6 months
  Adherence will be measured as the difference between the total hours medical device use from baseline to 3 months and from 3 months to 6 months (NightBalance SPT superior to PAP)

SECONDARY OUTCOMES:
Daytime Sleepiness | Baseline,3 months and 6 months
  Daytime sleepiness is measured using Epworth Sleepiness Scale (ESS). Epworth Sleepiness Scale (ESS), has a minimum value 0, maximum value 24 with higher values indicate worsening daytime sleepiness.
Impact of sleepiness on activities of daily living | Baseline,3 months and 6 months
  Impact of sleepiness on activities of daily living is measured using Functional Outcomes of Sleep Questionnaire (FOSQ). The FOSQ is a sleep related quality of life is measured across five dimensions; activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome. Each rate the difficulty of performing a given activity on a 4-point scale, min value 0, max value 4. Low scores indicate no difficulty, higher scores extreme difficulty.
Health related quality of life | Baseline,3 months and 6 months
  Health related quality of life is measured using EQ-5D at baseline and at the end of each 3 month treatment arm. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Responses are coded as single-digit numbers. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state with lower scores indicting worsening health status and higher values improved health status.
Fatigue | Baseline,3 months and 6 months
  Fatigue is measured using Pichot Fatigue Scale at baseline and at the end of each 3 month treatment arm. The Pichot Fatigue Scale is an 8 question survey in which is answered 0 to 4 with a maximum score of 32. A score above 22 reveals excessive fatigue, patients may suffer from inefficient sleep.
Quality of life utilizing SF-36 | Baseline,3 months and 6 months
  Quality of life is measured using SF-36 at baseline and at the end of each 3 month treatment arm. The 36-Item Short Form Health Survey (SF-36) is an indicator of overall health status. It has the following sections: Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health.
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. The lower scores mean more disability, and higher scores mean less disability.
Mean Disease Alleviation | 3 months and 6 months
  Mean Disease Alleviation is calculated using the AHI and adherence data at the end of each 3-month treatment arm 8. Adverse events are recorded at the end of each 3-month treatment arm
Health Economics and Resource Utilization | 3 months and 6 months
  Health Economics and Resource Utilization are assessed using healthcare utilization diary which is completed by patients during each 3-month treatment arm.

CONTACTS AND LOCATIONS:
Locations (18):
- France (6):
  - Centre Hospitalier Universitaire Angers, Angers
  - CHU Grenoble Alpes, Grenoble
  - Centre Hospitalier Universitaire Bordeaux, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Hôpital Universitaire Pitié - Salpêtrière (UPMC), Paris
  - Hopital Foch, Suresnes, Suresnes
- Germany (6):
  - Zentrum für Schlafmedizin Berlin, Berlin
  - Klinikum Rechts der Isar, München
  - Schlafmedizinisches Zentrum Regensburg, Regensburg
  - Praxis Dr. Holger Hein, Reinbek
  - Helios Kliniken, Schwerin
  - Hospital Bethanien Solingen, Solingen
- United Kingdom (6):
  - Royal Papworth Hospital, Cambridge
  - Royal infirmary of Edinburgh, Edinburgh
  - Prince Philip Hospital, Llanelli
  - Guy's and St Thomas' NHS Foundation Trust (GSTT), London
  - Royal Preston Hospital, Preston
  - North Tyneside General Hospital, Tyneside